CLINICAL TRIAL: NCT02856555
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety, Tolerability, and Efficacy of GS-0976 in Subjects With Nonalcoholic Steatohepatitis
Brief Title: Study to Evaluate Safety, Tolerability, and Efficacy of GS-0976 in Adults With Nonalcoholic Steatohepatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-426-3989
Record Dates: First submitted 2016-08-02; First posted 2016-08-05 (Estimated); Results first posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Nonalcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — firsocostat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Firsocostat 5 mg (Experimental): Participants will receive firsocostat 1 x 5 mg + 1 x placebo matched to firsocostat 5 mg + 2 x placebo matched to firsocostat 10 mg for 12 weeks.
  Interventions: Drug: Firsocostat; Drug: Placebo
- Firsocostat 20 mg (Experimental): Participants will receive firsocostat 2 X 10 mg + 2 x placebo matched to firsocostat 5 mg for 12 weeks.
  Interventions: Drug: Firsocostat; Drug: Placebo
- Placebo (Experimental): Participants will receive 2 x placebo matched to firsocostat 5 mg + 2 x placebo matched to firsocostat 10 mg for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Firsocostat — Capsules orally once daily.
  Other Names: GS-0976
  Arms: Firsocostat 20 mg; Firsocostat 5 mg
Drug: Placebo — Placebo matched to firsocostat orally once daily.

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of firsocostat in adults with nonalcoholic steatohepatitis (NASH).

ELIGIBILITY:
Key Inclusion Criteria:

* Meets all of the following conditions:

  * A clinical diagnosis of nonalcoholic fatty liver disease (NAFLD)
  * Screening magnetic resonance imaging - proton density fat fraction (MRI-PDFF) with ≥ 8% steatosis
  * Screening magnetic resonance elastography (MRE) with liver stiffness ≥ 2.5 kPa

    * OR
  * A historical liver biopsy consistent with NASH and non-cirrhotic fibrosis
* Platelet count ≥ 100,000/mm^3
* Creatinine Clearance (CLcr ) as calculated by the Cockcroft-Gault equation ≥ 60 ml/min

Key Exclusion Criteria:

* Pregnant or lactating females
* Alanine aminotransferase (ALT) > 5 x upper limit of the normal range (ULN)
* Other causes of liver disease including autoimmune, viral, and alcoholic liver disease
* Cirrhosis of the liver

  * Prior history of decompensated liver disease, including ascites, hepatic encephalopathy or variceal bleeding
* Body mass index (BMI) < 18 kg/m^2
* International normalized ratio (INR) > 1.2 unless on anticoagulant therapy
* Total bilirubin > 1 x ULN, except with diagnosis of Gilbert's syndrome

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2016-08-08 (Actual); Primary Completion 2017-07-18 (Actual); Study Completion 2017-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (30):
- United States (30):
  - Coronado, California
  - Foster City, California
  - Los Angeles, California
  - Rialto, California
  - San Diego, California
  - San Francisco, California
  - Miami, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Rochester, Minnesota
  - Kansas City, Missouri
  - New York, New York
  - Durham, North Carolina
  - Statesville, North Carolina
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Germantown, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Arlington, Texas
  - Live Oak, Texas
  - San Antonio, Texas
  - Murray, Utah
  - Falls Church, Virginia
  - Richmond, Virginia
  - Richland, Washington
  - Seattle, Washington

REFERENCES:
- [Result] Loomba R, Kayali Z, Noureddin M, Ruane P, Lawitz EJ, Gitlin N, Bennett M, Harting EJ, McColgan BJ, Myers RP, Subramanian GM, McHutchison JG, Middleton MS, Sirlin C, Lai M, Charlton M, Harrison SA. Acetyl-CoA carboxylase (ACC) inhibitor GS-0976 leads to significant improvements in MRI-PDFF in a Phase 2, randomized, placebo-controlled trial of patients with NASH. American Association for the Study of Liver Diseases Meeting; 2017; Washington, DC, USA.
- [Derived] Loomba R, Kayali Z, Noureddin M, Ruane P, Lawitz EJ, Bennett M, Wang L, Harting E, Tarrant JM, McColgan BJ, Chung C, Ray AS, Subramanian GM, Myers RP, Middleton MS, Lai M, Charlton M, Harrison SA. GS-0976 Reduces Hepatic Steatosis and Fibrosis Markers in Patients With Nonalcoholic Fatty Liver Disease. Gastroenterology. 2018 Nov;155(5):1463-1473.e6. doi: 10.1053/j.gastro.2018.07.027. Epub 2018 Jul 27. PMID 30059671
- [Derived] Lawitz EJ, Coste A, Poordad F, Alkhouri N, Loo N, McColgan BJ, Tarrant JM, Nguyen T, Han L, Chung C, Ray AS, McHutchison JG, Subramanian GM, Myers RP, Middleton MS, Sirlin C, Loomba R, Nyangau E, Fitch M, Li K, Hellerstein M. Acetyl-CoA Carboxylase Inhibitor GS-0976 for 12 Weeks Reduces Hepatic De Novo Lipogenesis and Steatosis in Patients With Nonalcoholic Steatohepatitis. Clin Gastroenterol Hepatol. 2018 Dec;16(12):1983-1991.e3. doi: 10.1016/j.cgh.2018.04.042. Epub 2018 Apr 26. PMID 29705265

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United States. The first participant was screened on 08 August 2016. The last study visit occurred on 18 July 2017.
Pre-assignment Details: 433 participants were screened.
Groups:
- Firsocostat 5 mg: Participants received firsocostat 1 x 5 mg + 1 x placebo matched to firsocostat 5 mg + 2 x placebo matched to firsocostat 10 mg capsules orally once daily for 12 weeks.
- Firsocostat 20 mg: Participants received firsocostat 2 x 10 mg + 2 x placebo matched to firsocostat 5 mg capsules orally once daily for 12 weeks.
- Placebo: Participants received 2 x placebo matched to firsocostat 5 mg + 2 x placebo matched to firsocostat 10 mg capsules orally once daily for 12 weeks.
Period: Overall Study
Arm/Group | Firsocostat 5 mg | Firsocostat 20 mg | Placebo
Started | 51 | 50 | 26
Completed | 46 | 46 | 26
Not Completed | 5 | 4 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 3 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — Randomized but Never Treated | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Firsocostat 5 mg | Firsocostat 20 mg | Placebo | Total
Number analyzed (Participants) | 51 | 49 | 26 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (11.6) | 54 (12.2) | 56 (9.6) | 54 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 33 | 19 | 82
  Male | 21 | 16 | 7 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 23 | 8 | 47
  Not Hispanic or Latino | 35 | 26 | 18 | 79
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1 | 0 | 1 | 2
  Race: Asian | 5 | 1 | 1 | 7
  Race: Black or African American | 3 | 2 | 1 | 6
  Race: White | 42 | 44 | 23 | 109
  Race: Others | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events
Time Frame: First Dose date up to last dose (Week 12) plus 30 days
Population: The Safety Analysis Set included participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Firsocostat 5 mg | Firsocostat 20 mg | Placebo
Number analyzed (Participants) | 51 | 49 | 26
percentage of participants | 70.6 | 71.4 | 61.5

ADVERSE EVENTS:
Time Frame: First Dose date up to last dose (Week 12) plus 30 days
Description: The Safety Analysis Set included participants who received at least 1 dose of study drug.
Arm/Group | Firsocostat 5 mg | Firsocostat 20 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/49 | 0/26
Serious Adverse Events (participants affected / at risk) | 2/51 | 2/49 | 0/26
Other Adverse Events (participants affected / at risk) | 26/51 | 29/49 | 11/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Firsocostat 5 mg (N=51) | Firsocostat 20 mg (N=49) | Placebo (N=26)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Firsocostat 5 mg (N=51) | Firsocostat 20 mg (N=49) | Placebo (N=26)
Nausea (Gastrointestinal disorders) | 4 | 7 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 6 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 5 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 4 | 1
Vomiting (Gastrointestinal disorders) | 1 | 5 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 2
Fatigue (General disorders) | 2 | 4 | 3
Chest discomfort (General disorders) | 0 | 0 | 2
Sinusitis (Infections and infestations) | 2 | 3 | 3
Influenza (Infections and infestations) | 0 | 5 | 1
Viral upper respiratory tract infection (Infections and infestations) | 3 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5 | 1 | 0
Headache (Nervous system disorders) | 5 | 4 | 1
Anxiety (Psychiatric disorders) | 3 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2016-12-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT02856555/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT02856555/SAP_001.pdf